CLINICAL TRIAL: NCT05550272
Title: Inventory of Hospitalizations in the Neonatal Period and Validation of the Early Maternity Discharge Protocol: Retrospective Observational Study
Brief Title: Hospitalizations in Neonatal Period and Early Discharge of Maternity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jourdan Laurélia, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2022PI110
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Hospitalization; Neonatal Period; Early Maternity Discharge; Risk Factor Readmission
Keywords: neonatal; readmission; early discharge maternity; causes of readmission

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
in the past 2 decades the number of early discharge of maternity is increasing. The aim of this study is to observe if an early maternity discharge increase the rate of hospitalization during the neonatal period.

All infants with maximum 28 days old who are hospitalized at the Hospital center of Nancy: through emergency unit of children's hospital or maternity, through intensive care unit of children's hospital.

ELIGIBILITY:
Inclusion Criteria:

* infants hospitalized maximum at the aged of 28 days (day 28 included)
* infants already discharged from maternity
* infants hospitalized in Hospital Center NANCY: at Children's
* informed by the study, parents did not refused to participate to the study

Exclusion Criteria:

* more than 28 days old
* infants transferred from maternity without discharge at home.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: hospitalized infants less than 28 days old at CHU Nancy hospital through the emergency service of children's hospital, through intensive care unit or through emergency unit of the maternity regional of Nancy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Age at maternity discharge | 1 month
  age in hours at the discharge of maternity

SECONDARY OUTCOMES:
Etiology of hospitalization | 1 month
  Description of the cause of the hospitalization
Jaundice risk factor | 1 month
  different risk factor of jaundice, jaundice and phototherapy
Risk factor of early neonatal bacterial infection | 1 month
  mother's and newborn's risk factor to determinate follow up
social environment at home, mother's parity | 1 month
  determined the environment of the newborn for a safety maternity discharge
pediatrics follow up | 1 month
  the follow up set up at home by the different medical stuff (pediatrician, family doctor, midwife